CLINICAL TRIAL: NCT05904483
Title: The Effects of Finger Puppet, Abeslang Puzzle, and Pinwheel on Pain and Anxiety in Children Aged 4-6 Years During Blood Sampling Procedures in Emergency Rooms: A Randomized Controlled Study
Brief Title: The Effects of Finger Puppet, Abeslang Puzzle, and Pinwheel on Pain and Anxiety During Blood Sampling Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Fatma Dinç, Principal Investigator, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-BRT-SBF-112234
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Pain, Acute; Anxiety; Child, Only
MeSH Terms: conditions — Acute Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pinwheel Group (Experimental): In the pinwheel group, a windmill made of colored cardboard is introduced to the children, and then they are asked to blow on the pinwheel during the blood sampling procedure.The blood sampling is terminated at the same time by blowing the pinwheel.
  Interventions: Other: PFA
- Finger Puppet Group (Experimental): In the finger puppet group, a finger puppet made of felt is introduced to the children, and they are told a story (Brave Little Rabbit) by the same researcher using the finger puppet.The blood sampling is terminated at the same time by reading story with finger puppet.
  Interventions: Other: PFA
- Abeslang Puzzle Group (Experimental): In the abeslang puzzle group, a puzzle made of colorful abeslang pieces with animal images (sheep, duck) is introduced to the children, and then they are asked to complete the puzzle using their non-dominant hand during the blood sampling procedure.The blood sampling is terminated at the same time by completing abeslang puzzle.
  Interventions: Other: PFA
- Control (No Intervention): Children in the control group are monitored during the blood sampling procedure if their informed consent is obtained by the researcher. They have the routine blood draw procedure, and do not receive any distraction techniques and other pharmacological interventions.

INTERVENTIONS:
Other: PFA — PFA
  Arms: Abeslang Puzzle Group; Finger Puppet Group; Pinwheel Group

SUMMARY:
Blood sampling is an invasive, diagnostic, and therapeutic procedure for children. The inability of preschool children to differentiate between reality and imagination and their belief in the power of their thoughts make it difficult for them to accept an invasive procedure. Distraction techniques are used to help children cope with pain and anxiety. The aim of this study is to compare the effects of finger puppet, abeslang puzzle, and pinwheel on pain and anxiety during blood sampling in preschool children presenting to the pediatric emergency department. This randomized controlled study used parallel trial design.

DETAILED DESCRIPTION:
The research hypotheses are as follows: H1: Children in the finger puppet group experience lower procedure-related pain than those in the control group. H2: Children in the pinwheel group experience lower procedure-related pain than those in the control group. H3: Children in the abeslang puzzle group experience lower procedure-related pain than those in the control group. H4: Children in the finger puppet group have lower anxiety than those in the control group. H5: Children in the pinwheel group have lower anxiety than those in the control group. H6: Children in the abeslang group have lower anxiety than those in the control group.

Methods:

This randomized controlled study plans to include children aged 4-6 years presenting to the pediatric emergency department of Bartın Maternity and Child Health Hospital. The study utilizes a parallel trial design, defining three different intervention groups (pinwheel, abeslang puzzle, finger puppet) and a control group (standard care). An independent statistician (www.randomize.org) allocates participants to groups using a randomization method according to sampling criteria. Since there is no similar study about the effects of finger puppet, abeslang puzzle, and pinwheel on pain and anxiety during blood sampling in children, the study aims for a medium effect size (0.25) to determine the sample size (Cohen, 2013). Considering a medium effect size (f: 0.25), a power of 80% (1 - β error), and a confidence level of 95% (α error), the sample of the study should include 180 children (G*Power 3.1.9.7) (Faul, 2014). Considering potential data losses, the sample size is increased by 10%, resulting in 200 children with 50 children in each group. Children and their parents are informed about the study, and after obtaining their consent, they are assigned to their respective groups.

A standard approach is applied to all pediatric patients, which includes providing information about the procedure, introducing the nurse, selecting the intervention area together, having the parent present during the procedure, and engaging in conversation with the child. No additional intervention is applied to children in the control group, and after obtaining their parental consent, they are observed during the procedure.

In the finger puppet group, a finger puppet made of felt is introduced to the selected child, and a story (Brave Little Rabbit) is told using the finger puppet. The finger puppet is wiped with a disinfectant before and after the intervention.

In the abeslang puzzle group, a puzzle made of colorful abeslang pieces with animal images (sheep, duck) is introduced to the selected child, and then the child is asked to complete the puzzle using their non-dominant hand, while the blood sampling procedure is being performed. Each child in the abeslang puzzle group receives the same number of puzzle pieces with the same design.

In the pinwheel group, a windmill made of colored cardboard is introduced to the selected child, and then the child is asked to blow on the pinwheel during the blood sampling procedure. The pinwheel is wiped with a disinfectant before and after the intervention.

All blood sampling procedures are performed by the same nurse, and the same researcher is present during all interventions.

Research data is collected by the following data collection forms:

Personal Information Form: The form consists of 4 questions in total, including age, gender, presence of previous injection experience, and number of previous injection experience.

Wong-Baker FACES (WB-FACES) Pain Rating Scale: This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10.

The Children's Anxiety Meter (CAM). This scale assesses children's anxiety in clinical settings and uses before medical procedures. Children are asked to mark how they feel "right now" to measure state anxiety (CAM-S). Scores range from 0 to 10. It validated at children aged 4-10 years during an intravenous procedure.

ELIGIBILITY:
Inclusion Criteria:

* Being between 4-6 years old
* Referring to the pediatric emergency department
* Having consent and approval from the parent and child to participate in the study
* Having a necessity for blood testing in the child.

Exclusion Criteria:

* Having visual, hearing, or speech impairment
* Having chronic or genetic diseases
* Having intellectual disability
* Having a history of sedative, narcotic, or analgesic drug use within the past 24 hours
* Having inflammatory diseases
* Being classified under the red triage category
* Unwilling to participate in the study.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
The level of pain during blood sampling is evaluated using the Wong-Baker FACES Pain Rating Scale | during the procedure
  This scale is used to assess the severity of pain in children aged 3 years and above. This numerical rating scale ranges from 0 to 10, indicating emotions ranging from no pain/very happy (0) to crying/hurts worst (10). Higher scores indicate a lower pain tolerance. In this study, this scale is evaluated using personal reports and records from children, their parents, the researcher, and the nurse after the blood sampling procedure.

SECONDARY OUTCOMES:
The level of anxiety is evaluated using the Children Anxiety Meter-State | during the procedure
  The Children's Anxiety Meter (CAM-S) assesses children's anxiety in clinical settings and is used prior to medical procedures. The CAM is drawn like a thermometer with a bulb at the bottom and contains horizontal lines at intervals going upwards. Scale scores range from 0 to 10, where higher values represent higher anxiety. Personal reports and records from children, their parents, the researcher, and the nurse, who are asked to mark the scale with a pen, are used to assess the anxiety levels of children regarding blood sampling before and after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Dinç, PhD Student, Principal Investigator — Bartın Unıversity
Locations (1):
- Fatma Dinç, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Dinc F, Kurt A, Gunes San E. The effect of three different methods on pain and anxiety in children during blood sampling procedure in pediatric emergency department: Finger puppet, abeslang puzzle, pinwheel. J Pediatr Nurs. 2024 Nov-Dec;79:e203-e212. doi: 10.1016/j.pedn.2024.10.023. Epub 2024 Oct 24. PMID 39448323